CLINICAL TRIAL: NCT02448823
Title: Evaluating Demand Generation (Stylish Man, Stylish Living) for HIV Prevention/Family Planning Services, Rakai, Uganda
Brief Title: Evaluating Demand Generation (Stylish Man , Stylish Living) for HIV Prevention/Family Planning Services, Rakai, Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Rakai Health Sciences Program (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AI114438; R01AI114438 (NIH); NCT02476071 (obsolete NCT alias)
Record Dates: First submitted 2014-09-23; First posted 2015-05-20 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2019-04

CONDITIONS: HIV
Keywords: HIV; combined prevention; demand generation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stylish Events and Mass Media (Experimental): Mass Media (radio, posters) and annual Stylish Man/Stylish Living Event (SMLEvent), a multimedia event promoting CHP.
  Interventions: Other: Mass media and Stylish Events
- Control arm: mass media only (Active Comparator): Mass media
  Interventions: Other: Mass Media

INTERVENTIONS:
Other: Mass media and Stylish Events — 1. Mass media (MM): Radio broadcasts, dramatized dialogues, interviews with opinion leaders and satisfied clients . Posters.
  2. "Stylish Man/Living Event" (SMLEvent) community mobilization/service provision. SMLEvent activities. Messages on how CHP (including behaviors such as sexual risk reduction) can make men and women feel more in control of their lives, less stressed, and more "Stylish" are interwoven through the mobilization.
  The Stylish Man Van (SMV) accompanies the SMLEvent. The Van includes multimedia and health mobilizers who insert HIV prevention messages, testimonials by satisfied CHP "customers" and where appropriate their spouses.
  Arms: Stylish Events and Mass Media
Other: Mass Media — 1. Mass media (MM): Radio broadcasts, dramatized dialogues, interviews with opinion leaders and satisfied clients . Posters.
  Arms: Control arm: mass media only

SUMMARY:
The study tests a novel demand generation strategy, "Stylish Man/Stylish Living", to increase uptake of Combined HIV Prevention (CHP) in Rakai, Uganda. CHP includes safe voluntary medical male circumcision (VMMC), antiretroviral therapy (ART), and behavioral interventions. With President's Emergency Fund for AIDS Relief (PEPFAR) funds, the Rakai Health Sciences Program (RHSP) provides CHP in Rakai District, Uganda. Our ongoing 54 village Rakai Community Cohort Study (RCCS), with community HIV prevalence ranging from 6% to 42%, provides longitudinal data on rates of CHP coverage and on HIV incidence. There is preliminary evidence that CHP is reducing HIV incidence in Rakai, but CHP coverage remains suboptimal, particularly in men. Data suggest that CHP supply is not the limiting factor, but that there is a "deficit in demand".

Based on extensive qualitative research, we developed an innovative male-focused CHP demand generation strategy, the "Stylish Man/Stylish Living Program" (SMLP) which is male-friendly without excluding women. SMLP strives to "demedicalize" CHP by de-emphasizing health-focused messages and instead stressing "taking charge of your life". It has two related elements: (1) mass media (MM) via radio and posters; and (2) community-level mobilization via the "Stylish Man/Stylish Living Event" (SMLEvent) which includes CHP promotion through multimedia (the Stylish Van, videos, music, health promoters) and immediate access to services (mobile camps which offer VMMC camps, HIV testing and counseling services, referral for ART, and contraceptive services). In this study, the investigators will conduct a 4.5 year cluster randomized trial of MM/mobile service camps+SMLEvents (intervention arm) compared to MM/mobile service camps conducted without SMLEvents (control), in 25 RCCS communities per arm aggregated into ~10 clusters per arm (50 communities in all). The primary outcome will be intent-to-treat community-level rates of CHP coverage by arm, and service statistics on use of mobile camp services by arm. The investigators will also monitor rates of key behaviors and HIV incidence, and compare them between arms and to rates observed in communities in each arm prior to study initiation (secondary outcomes).

DETAILED DESCRIPTION:
Assessment strategy:

We propose a pragmatic cluster-randomized trial of the effects of MM/mobile service camps+SMLEvent (intervention) versus MM/mobile service camps without SMLEvents (control) on CHP coverage and on usage of mobile camp services by arm. In addition, RCCS data from before and after trial initiation will provide data on trends in CHP coverage, HIV incidence and key behaviors in both arms before and during the trial. The "pragmatic" approach allows modification of the SMLP components based on feedback and iterative assessments, as would be the case in normal program practice.

Cluster randomized trial component:

* 50 Rakai Community Cohort Study (RCCS) communities will be divided into ~20 clusters of 2-3 villages in close geographic proximity per arm. The total population of all 50 communities is ~18,000, of whom we estimate approximately 15,000 will be interviewed via the RCCS as a component of intervention evaluation. The clusters will be stratified by community characteristics (e.g., fishing villages, main road hubs, agrarian villages), and randomized within strata.

Intervention arm: ~ ten clusters will be randomly assigned to receive the SMLEvent activities once ~ annually for 3 cycles in addition to the ongoing district-wide MM. The SMLEvents will include the community mobilization as described above, carried out in conjunction with mobile service camps conducted at the time of the SMLEvent.

The other ~10 clusters (control arm) will be exposed to MM for 3 cycles but will not receive SMLEvents. All control communities will be offered all CHP services via RHSP/Ministry of Health (MOH) mobile clinics conducted for the same 3 cycles in conjunction with RCCS survey rounds.

Both intervention and control arm clusters will continue to have year-round access to existing MOH/RHSP clinic CHP services. Services in both arms will be offered per Uganda Centers for Disease Control and Prevention (CDC) PEPFAR guidelines. Both arms will thus have equivalent access to CHP.

Pre-post component:

The MM campaign on radio which covers a large proportion of the population of Rakai cannot be randomized. However, the RCCS provides longitudinal information on population-level rates of HIV care/ART for the general population and for pregnant women (p-MTCT), VMMC and family planning, as well as data on behaviors (condom use, numbers of partners, etc…) and HIV incidence, since 1994. Thus, within control arm communities, we have data required to determine what proportion of the population are exposed to the mass media, and whether the MM is associated with increased demand and among which population subgroups. The rate of service uptake in the RCCS has essentially plateaued for over the past 3 RCCS rounds, so an upward inflection following MM startup will suggest program effects. We will also conduct a pre-post comparison in the SMLEvent+MM arm.

As described below, we will add questions to the RCCS to enhance the SMP evaluation. CHP uptake will also be assessed with mobile camp service statistics in both study arms.

Methods of data collection:

1. Annual RCCS community surveillance surveys, among all consenting individuals aged 15-49 in the 50 RCCS communities (aggregated into ~10 clusters per trial arm).

   The RCCS will continue to collect detailed data on sociodemographics, behaviors (including numbers and types of partners, condom use with each, whether the partner is from within the community or another geographic setting), egocentric sexual network, pregnancy since the last RCCS survey round, health status and use of HCT, condoms, ART, P-MTCT, and VMC. We will add a module in the RCCS to evaluate exposure to the SMLP (mass media, SMLEvent), perceptions of components of the SMLP (both positive and negative), perceptions of different CHP services and the degree to which they are acceptable within the respondent's family, peer group and community; whether the respondent has had conversations with partners, family and/or peers about any CHP services; whether an individual accepted any service or adopted any self-reported behavioral change as a result of the campaign, and if so, what was (were) the main influence(s) (i.e., information, found out peers were using services, friends or spouses encouraged uptake as a result of the campaign, easier access to the service, etc….. ) HIV testing will be conducted at each RCCS survey round, using a three rapid test algorithm, with EIA and/or PCR confirmation of all newly identified HIV+ in-migrants and all new seroconverters. Serum samples from the RCCS will be archived at -800C for future studies such as community viral load, under future grants. Women will be asked about pregnancy status; those who are uncertain will be offered a urinary hCG pregnancy test (this is offered routinely in the RCCS). Pregnant HIV+ women will be referred for p-MTCT.

   Since the RCCS routinely collects serum for HIV testing and CD4, we will track HIV incidence, and immunologic status through the RCCS, complementing the clinic-based evaluation described below.
2. Process data:

   Records will be kept of each SMLP activity: radio spots and interviews, scheduling of SMLEvent activities, etc. SMLEvent process data will include estimates of the number of participants each day, with photos taken to assist with the count. Approximately 12 short anonymous "spot interviews" will be conducted daily at the SMLEvent site daily with younger and older men and women, to gauge interest in the activities, positive and negative perceptions, and suggestions for improvement.
3. Clinic-based evaluation:

In both study arms, we will collect service statistics from the mobile CHP camps (mobile camps plus SMLEvents in the intervention arm, and stand-alone service camps in the control arm)by services and referrals provided, client's age, gender, venue and date. Please note: the sand-alone mobile camps int he control arm will be announced to the community approximately two weeks prior to their occurrance, in order to ensure potential clients are aware of them; however, this notification will not include the multimedia and community mobilization associated with the SMLEvents. (Client medical records will include the individual's name, but will be retained separately from research records.) Clients will be asked what motivated them to accept a service (some SMLP component, other people were getting services, encouragement from someone influenced by the SMLP, factors unrelated to the SMLP, etc…) We will track whether persons referred for HIV care/ART present to our HIV clinics (and conversely, we will ask about clinic attendance during each RCCS survey rounds). Routine HIV clinic data collection includes tracking of visits, questions on adherence, and CD4 cell count every 6 months. PEPFAR does not currently fund HIV viral load, but samples from the RHSP/MOH clinics are tested for viral load annually with International Center for Excellence in Research (ICER) funds. These data will complement the RCCS data, providing a comprehensive indication of ART coverage and long term treatment outcomes.

Cost data:

We do not propose a formal cost benefit analysis. However, the cost of the campaign will be closely tracked (cost of each radio spot, personnel/materials for the SMLEvent, fuel, administrative and support costs, additional cost to PEPFAR of extended evening service hours, etc…). The focus will be on service-related costs, with research outlays tracked separately. We will compare overall costs per unit ART, VMC and p-MTCT coverage, in the intervention versus the control arm and in relation to PEPFAR costs per client to date.

ELIGIBILITY:
Please note: the question above ("accepts health volunteers") is not really applicable to this community randomized trial. We are not enrolling anyone into the trial, and we are not testing any individual level interventions: by definition, all community members can be exposed to the messages on radio and posters, and anyone can come to the Stylish Man/Stylish Living event. We will interview approximately 15,000 persons in the study communities about their exposure to the Stylish Program and regarding their use of CHP services, as part of our ongoing, longitudinal Rakai Community Cohort Study (RCCS), in which we have already been asking about use of CHP services since they were first introduced, starting in approximately 2004. However, being interviewed in the RCCS is in no way dependent on having been exposed to the Stylish Program. We will also collect service statistics at mobile CHP service delivery camps in both arms. However, we already routinely conduct such camps throughout RCCS communities and offer standard-of-care CHP services. The one difference will be that in the intervention arm communities, community mobilization and multimedia information will be provided via the SMLEvents.

Inclusion Criteria:

* Residents aged 18-49 years in the 50 communities. (Please note: this is a community-randomized trial)

Exclusion Criteria:

* All community residents may attend the events and by definition, will be exposed to mass media. However, only persons aged 18-49 who sign or fingerprint a written informed consent will be interviewed in the RCCS as part of the evaluation nested within the RCCS.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17386 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Community level uptake of selected combined HIV prevention services (HIV testing and counseling services, VMMC, referral for HIV care/ART, family planning. | 5 year study
  Clients will be asked what motivated them to accept a service (some SMLP component, other people were getting services, encouragement from someone influenced by the SMLP, factors unrelated to the SMLP, etc…) We will track whether persons referred for HIV care/ART present to our HIV clinics (and conversely, we will ask about clinic attendance during each RCCS survey rounds). Routine HIV clinic data collection includes tracking of visits, questions on adherence, and CD4 cell count every 6 months
Service statics in mobile service camps in each study arm | 5 year study
  Data will be recorded regarding the numbers and characteristics of clients accepting HIV counseling and testing services, VMMC, referral for ART, and family planning, by age, gender and community.

SECONDARY OUTCOMES:
Selected HIV risk behaviors and HIV incidence | 5 year study
  We will assess rates of key behaviors and HIV incidence over time; these are secondary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Wawer, MD, MHSc, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Rakai Health Sciences Program, Kalisizo, Rakai District, Uganda